CLINICAL TRIAL: NCT04607057
Title: The Effect of Postoperative Supplemental Parenteral Nutrition (SPN) in Gastric Cancer Patients Who Underwent Gastrectomy: A Multicenter Prospective Randomized Controlled Trial
Brief Title: Supplemental Parenteral Nutrition During Postgastrectomy in Nutritionally at Risk Patient
Acronym: SUPPORT
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Hyuk-Joon Lee, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-2005-159-1126
Record Dates: First submitted 2020-10-12; First posted 2020-10-28 (Actual); Last update posted 2021-09-24 (Actual); Status verified 2021-09

CONDITIONS: Gastric Cancer; Gastrectomy; Malnutrition
Keywords: Gastric cancer; Postgastrectomy; Malnutrition; Supplemental; Parenteral nutrition
MeSH Terms: conditions — Stomach Neoplasms; Malnutrition; Hyperphagia | interventions — Parenteral Nutrition Solutions

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Arm A) (Experimental): Preparation of parenteral nutrition (PN): Among winuf(1820cc for central vein, 1,450cc for peripheral vein), smofkabaven(986cc for central vein, 1206cc for peripheral vein), and nutriplex(1875cc for central vein, 1,250cc for peripheral vein) Amount of PN: Total energy expenditure (TEE) of the patients will be calculated with Harris-Benedict Equation, activity factor, and stress factor. The amount of calorie from oral intake will be subtracted from TEE then the remainder will be provided through PN.
  Route of PN Injection: PICC (percutaneously-inserted central catheter) will be secured for PN for the central vein. PN for the peripheral vein will be injected directly through peripheral superficial vein.
  * Day0 : fasting(NPO) + crystalloid fluid
  * POD#1 : Keep fasting, then start sips of water in the evening + crystalloid fluid
  * POD#2 : Semifluid diet (SFD) + crystalloid fluid
  * POD#3 : Semifluid diet (SFD) + PN
  * POD#4-7: Soft blended diet (SBD) + PN
  Interventions: Drug: Parenteral Nutrition Solutions
- control group (Arm B) (No Intervention): * Day0 : fasting(NPO) + crystalloid fluid
  * POD#1 : Keep fasting, then start sips of water in the evening + crystalloid fluid
  * POD#2 : Semifluid diet (SFD) + dextrose 5% water
  * POD#3 : Semifluid diet (SFD) + dextrose 5% water
  * POD#4-7: Soft blended diet (SBD)

INTERVENTIONS:
Drug: Parenteral Nutrition Solutions — * Day0 : fasting(NPO) + crystalloid fluid
  * POD#1 : Keep fasting, then start sips of water in the evening + crystalloid fluid
  * POD#2 : Semifluid diet (SFD) + crystalloid fluid
  * POD#3 : Semifluid diet (SFD) + PN
  * POD#4-7: Soft blended diet (SBD) + PN
  Arms: experimental group (Arm A)

SUMMARY:
* If a patient undergoes gastrectomy, which is a kind of major abdominal operation, he/she loses more than 5% of his/her body weight in 2 months after surgery. This point is one of the criteria of 'risk of malnutrition' according to Nutrition Risk Screening (NRS 2002) and the patient who corresponds to this criterion needs nutritional support.
* According to Nutrition Risk Screening (NRS 2002), moderate malnutrition is defined as the state that the patient orally intakes 25~50% of recommended requirements; severe malnutrition is less than 25%.
* Meanwhile, when oral nutrition support was provided to patients after gastric cancer surgery, the patients' average daily intake during the first three months was about a half of the recommended requirements.

  * Putting together the facts i) that the patient underwent major abdominal operation, ii) that the weight loss rate exceeded 5% for two months, iii) that the average daily intake of patients during the first three months was about half of the recommended amount, the patients are eligible to be classified as a group who require nutritional support according to NRS 2002.

Therefore, it is intended to verify the efficacy and safety of supplemental parenteral nutrition by comparing Arm A, who are provided oral intake with supplemental parenteral nutrition, Arm B, who are provided oral intake only after curative gastric cancer surgery.

DETAILED DESCRIPTION:
With at least 5 days of supplemental parenteral nutrition, we expect minimized body weight loss, favorable blood test result, eligibility for chemotherapy compliance, increased quality of life (QoL), decreased infection rate, decreased hospital stay, and decreased mortality.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who will undergo curative gastric cancer surgery (total gastrectomy, distal gastrectomy, proximal gastrectomy, and pylorus-preserving gastrectomy)
2. A Malnourished patient who meets one or more of the following:

   * BMI ≤ 20.5 kg/m2: BMI will be measured 1 day before surgery
   * Rapid weight loss (decreased by more than 5% in 2 months)
3. Patients over 18 years of age
4. Patients who are expected to receive PN for more than five days after surgery
5. Patients who are able to eat orally, but cannot fulfill the recommened calorie requirement by oral intake alone.

Exclusion Criteria:

1. In case that the patients have already provided parenteral nutrition prior to the consent of the study (oral diet prior to consent has nothing to do with study)
2. In case that the patients need tube feeding
3. Patients who are contraindicated to parenteral nutrition: heart failure (if the patient has current symptoms or receiving heart failure treatment, if ejection fraction(EF) was less than 40% in preoperative echocardiogram), Child-Pugh score C, renal failure (patient with 50% increased creatinine more than upper normal limit, patients currently undergoing renal replacement therapy), and pulmonary edema (appropriate chest X-ray signs for pulmonary edema), and the patient who suffered from allergie reaction to parenteral nutrition solutions.
4. Patients who are not easily able to obtain venous pathways or are vulnerable to side effects due to venous pathways (e.g. increased infection risk due to immunosupressant status)
5. Vulnerable subject (those who lack the decision making ability, pregnant women, or women who are planning to conceive)
6. Other patients whom the investigator has determined to be inappropriate to participate in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 224 (Estimated)
Dates: Start 2020-12-22 (Actual); Primary Completion 2022-10-30 (Estimated); Study Completion 2022-10-30 (Estimated)

PRIMARY OUTCOMES:
Total amount of calorie provision during hospitalization | discharge day (POD#8; postoperative day 8)
  kcal (kilocalorie)
Body weight change for 2 months after surgery | Outpatient (visit 2: 2 months ± 14 days after surgery)
  kg (kilogram)

SECONDARY OUTCOMES:
Body weight and fat free mass changes | Body weight: through study completion / Fat free mass: through study completion, an average of 1 year
  kg (kilogram)
Changes in blood test indicators : Hb | through study completion, an average of 1 year
  Complete blood count : Hb (hemoglobin) : g/dl
Changes in blood test indicators : WBC | through study completion, an average of 1 year
  Complete blood count : WBC (white blood cell) : cells/mm3
Changes in blood test indicators : lymphocyte | through study completion, an average of 1 year
  Complete blood count : lymphocyte (%)
Changes in blood test indicators : TLC | through study completion, an average of 1 year
  Complete blood count : TLC (total lymphocyte count) : cells/mm3
Changes in blood test indicators : total cholesterol | through study completion, an average of 1 year
  Blood chemistry : total cholesterol (mg/dl)
Changes in blood test indicators : total protein | through study completion, an average of 1 year
  Blood chemistry : total protein (g/dl)
Changes in blood test indicators : albumin | through study completion, an average of 1 year
  Blood chemistry : albumin (g/dl)
Changes in blood test indicators : AST | through study completion, an average of 1 year
  Blood chemistry : AST (aspartate aminotransferase) : IU/L
Changes in blood test indicators : ALT | through study completion, an average of 1 year
  Blood chemistry : ALT (alanine aminotransferase) : IU/L
Changes in blood test indicators : CRP | through study completion, an average of 1 year
  Blood chemistry : CRP (C-reactive protein) : mg/dl
Changes in serum cytokines | approximately up to 2 weeks
  ng/ml
Probability for chemotherapy : ECOG performance status | through study completion, an average of 1 year
  ECOG(Eastern Cooperative Oncology Group) performance status: 0~5 (higher scores mean a worse outcome) 0 : Fully active, able to carry on all pre-disease performance without restriction 5 : Death
Probability for chemotherapy : ASA score | through study completion, an average of 1 year
  ASA(American Society of Anaesthesiologists) score : 1~6 (higher scores mean a worse outcome)
  1 : A normal healthy patient 6 : A declared brain-dead patient whose organs are being removed for donor purposes
QoL : EORTC QLQ-C30 | through study completion, an average of 1 year
  EORTC QLQ-C30 (European Organization for Research and Treatment of Cancer Quality of Life Questionnaire - Core 30) : EORTC QLQ-C30 Scoring Manual (Fayers et al., 2001).
QoL : EORTC QLQ-STO22 | through study completion, an average of 1 year
  EORTC QLQ-STO22 (European Organization for Research and Treatment of Cancer Quality of Life Questionnaire - Stomach 22) : Clinical and psychometric validation of a questionnaire module, the EORTC QLQ-STO 22, to assess quality of life in patients with gastric cancer (J.M Blazeby el al. 2004).
QoL : SF-36 | through study completion, an average of 1 year
  SF-36 (36-Item Short Form Health Survey) : 0~100 (higher scores mean a worse outcome)
Infection rate | During the hospitalization (approximately up to 2 weeks)
  proportion
Total days of hospitalization | at Discharge Day (POD#8; postoperative day 8)
  day
Mortality rate | through study completion, an average of 1 year
  proportion

CONTACTS AND LOCATIONS:
Overall Officials: Hyuk-Joon Lee, Professor, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No
Sharing the specific individual participant data sets is not mandatory.

REFERENCES:
- [Background] Scholmerich J. Postgastrectomy syndromes--diagnosis and treatment. Best Pract Res Clin Gastroenterol. 2004 Oct;18(5):917-33. doi: 10.1016/j.bpg.2004.08.003. PMID 15494286
- [Background] Pedrazzani C, Marrelli D, Rampone B, De Stefano A, Corso G, Fotia G, Pinto E, Roviello F. Postoperative complications and functional results after subtotal gastrectomy with Billroth II reconstruction for primary gastric cancer. Dig Dis Sci. 2007 Aug;52(8):1757-63. doi: 10.1007/s10620-006-9655-6. Epub 2007 Apr 3. PMID 17404848
- [Background] Jee SH, Sull JW, Park J, Lee SY, Ohrr H, Guallar E, Samet JM. Body-mass index and mortality in Korean men and women. N Engl J Med. 2006 Aug 24;355(8):779-87. doi: 10.1056/NEJMoa054017. Epub 2006 Aug 22. PMID 16926276
- [Background] Migita K, Takayama T, Saeki K, Matsumoto S, Wakatsuki K, Enomoto K, Tanaka T, Ito M, Kurumatani N, Nakajima Y. The prognostic nutritional index predicts long-term outcomes of gastric cancer patients independent of tumor stage. Ann Surg Oncol. 2013 Aug;20(8):2647-54. doi: 10.1245/s10434-013-2926-5. Epub 2013 Mar 6. PMID 23463091
- [Background] Aoyama T, Yoshikawa T, Shirai J, Hayashi T, Yamada T, Tsuchida K, Hasegawa S, Cho H, Yukawa N, Oshima T, Rino Y, Masuda M, Tsuburaya A. Body weight loss after surgery is an independent risk factor for continuation of S-1 adjuvant chemotherapy for gastric cancer. Ann Surg Oncol. 2013 Jun;20(6):2000-6. doi: 10.1245/s10434-012-2776-6. Epub 2012 Dec 16. PMID 23242818
- [Background] Aoyama T, Sato T, Maezawa Y, Kano K, Hayashi T, Yamada T, Yukawa N, Oshima T, Rino Y, Masuda M, Ogata T, Cho H, Yoshikawa T. Postoperative weight loss leads to poor survival through poor S-1 efficacy in patients with stage II/III gastric cancer. Int J Clin Oncol. 2017 Jun;22(3):476-483. doi: 10.1007/s10147-017-1089-y. Epub 2017 Feb 7. PMID 28176023
- [Background] Beattie AH, Prach AT, Baxter JP, Pennington CR. A randomised controlled trial evaluating the use of enteral nutritional supplements postoperatively in malnourished surgical patients. Gut. 2000 Jun;46(6):813-8. doi: 10.1136/gut.46.6.813. PMID 10807893
- [Background] Smedley F, Bowling T, James M, Stokes E, Goodger C, O'Connor O, Oldale C, Jones P, Silk D. Randomized clinical trial of the effects of preoperative and postoperative oral nutritional supplements on clinical course and cost of care. Br J Surg. 2004 Aug;91(8):983-90. doi: 10.1002/bjs.4578. PMID 15286958
- [Background] Kong SH, Lee HJ, Na JR, Kim WG, Han DS, Park SH, Hong H, Choi Y, Ahn HS, Suh YS, Yang HK. Effect of perioperative oral nutritional supplementation in malnourished patients who undergo gastrectomy: A prospective randomized trial. Surgery. 2018 Dec;164(6):1263-1270. doi: 10.1016/j.surg.2018.05.017. Epub 2018 Jul 25. PMID 30055788
- [Background] Harvey SE, Parrott F, Harrison DA, Bear DE, Segaran E, Beale R, Bellingan G, Leonard R, Mythen MG, Rowan KM; CALORIES Trial Investigators. Trial of the route of early nutritional support in critically ill adults. N Engl J Med. 2014 Oct 30;371(18):1673-84. doi: 10.1056/NEJMoa1409860. Epub 2014 Oct 1. PMID 25271389
- [Background] Kong SH, Park JS, Lee IK, Ryu SW, Park YK, Yang HK, Han SU, Yoon KY, Jeong SY, Jeong MR, Hwang DW, Suh YS, Yoon YS, Seo KW, Park JW, Byun CS, Hur H, Won H, Choi Y, Lee HJ. Postoperative oral nutritional supplementation after major gastrointestinal surgery: a randomized controlled clinical trial. Asia Pac J Clin Nutr. 2017;26(5):811-819. doi: 10.6133/apjcn.112016.02. PMID 28802290
- [Background] Kondrup J, Rasmussen HH, Hamberg O, Stanga Z; Ad Hoc ESPEN Working Group. Nutritional risk screening (NRS 2002): a new method based on an analysis of controlled clinical trials. Clin Nutr. 2003 Jun;22(3):321-36. doi: 10.1016/s0261-5614(02)00214-5. PMID 12765673
- [Background] Kobayashi D, Ishigure K, Mochizuki Y, Nakayama H, Sakai M, Ito S, Kojima H, Kajikawa M, Ando M, Kodera Y. Multi-institutional prospective feasibility study to explore tolerability and efficacy of oral nutritional supplements for patients with gastric cancer undergoing gastrectomy (CCOG1301). Gastric Cancer. 2017 Jul;20(4):718-727. doi: 10.1007/s10120-016-0668-3. Epub 2016 Nov 24. PMID 27885538
- [Background] Russell MK, Wischmeyer PE. Supplemental Parenteral Nutrition: Review of the Literature and Current Nutrition Guidelines. Nutr Clin Pract. 2018 Jun;33(3):359-369. doi: 10.1002/ncp.10096. PMID 29878557
- [Background] Cahill NE, Dhaliwal R, Day AG, Jiang X, Heyland DK. Nutrition therapy in the critical care setting: what is "best achievable" practice? An international multicenter observational study. Crit Care Med. 2010 Feb;38(2):395-401. doi: 10.1097/CCM.0b013e3181c0263d. PMID 19851094
- [Background] Berger MM, Pantet O, Jacquelin-Ravel N, Charriere M, Schmidt S, Becce F, Audran R, Spertini F, Tappy L, Pichard C. Supplemental parenteral nutrition improves immunity with unchanged carbohydrate and protein metabolism in critically ill patients: The SPN2 randomized tracer study. Clin Nutr. 2019 Oct;38(5):2408-2416. doi: 10.1016/j.clnu.2018.10.023. Epub 2018 Nov 5. PMID 30448193
- [Background] Alberda C, Gramlich L, Jones N, Jeejeebhoy K, Day AG, Dhaliwal R, Heyland DK. The relationship between nutritional intake and clinical outcomes in critically ill patients: results of an international multicenter observational study. Intensive Care Med. 2009 Oct;35(10):1728-37. doi: 10.1007/s00134-009-1567-4. Epub 2009 Jul 2. PMID 19572118
- [Background] Compher C, Chittams J, Sammarco T, Nicolo M, Heyland DK. Greater Protein and Energy Intake May Be Associated With Improved Mortality in Higher Risk Critically Ill Patients: A Multicenter, Multinational Observational Study. Crit Care Med. 2017 Feb;45(2):156-163. doi: 10.1097/CCM.0000000000002083. PMID 28098623
- [Background] Heidegger CP, Berger MM, Graf S, Zingg W, Darmon P, Costanza MC, Thibault R, Pichard C. Optimisation of energy provision with supplemental parenteral nutrition in critically ill patients: a randomised controlled clinical trial. Lancet. 2013 Feb 2;381(9864):385-93. doi: 10.1016/S0140-6736(12)61351-8. Epub 2012 Dec 3. PMID 23218813
- [Background] Casaer MP, Mesotten D, Hermans G, Wouters PJ, Schetz M, Meyfroidt G, Van Cromphaut S, Ingels C, Meersseman P, Muller J, Vlasselaers D, Debaveye Y, Desmet L, Dubois J, Van Assche A, Vanderheyden S, Wilmer A, Van den Berghe G. Early versus late parenteral nutrition in critically ill adults. N Engl J Med. 2011 Aug 11;365(6):506-17. doi: 10.1056/NEJMoa1102662. Epub 2011 Jun 29. PMID 21714640
- [Background] Ridley EJ, Davies AR, Parke R, Bailey M, McArthur C, Gillanders L, Cooper DJ, McGuinness S; Supplemental Parenteral Nutrition Clinical Investigators. Supplemental parenteral nutrition versus usual care in critically ill adults: a pilot randomized controlled study. Crit Care. 2018 Jan 23;22(1):12. doi: 10.1186/s13054-018-1939-7. PMID 29361959
- [Background] Wu W, Zhong M, Zhu DM, Song JQ, Huang JF, Wang Q, Tan LJ. Effect of Early Full-Calorie Nutrition Support Following Esophagectomy: A Randomized Controlled Trial. JPEN J Parenter Enteral Nutr. 2017 Sep;41(7):1146-1154. doi: 10.1177/0148607116651509. Epub 2016 May 20. PMID 27208039
- [Background] Bai H, Li Z, Meng Y, Yu Y, Zhang H, Shen D, Chen L. Effects of parenteral omega-3 fatty acid supplementation in postoperative gastrointestinal cancer on immune function and length of hospital stay: a systematic review and meta-analysis. Asia Pac J Clin Nutr. 2018;27(1):121-128. doi: 10.6133/apjcn.022017.19. PMID 29222889
- [Background] Kim YG, Kong SH, Oh SY, Lee KG, Suh YS, Yang JY, Choi J, Kim SG, Kim JS, Kim WH, Lee HJ, Yang HK. Effects of screening on gastric cancer management: comparative analysis of the results in 2006 and in 2011. J Gastric Cancer. 2014 Jun;14(2):129-34. doi: 10.5230/jgc.2014.14.2.129. Epub 2014 Jun 30. PMID 25061541
- [Background] Visser M, Pahor M, Taaffe DR, Goodpaster BH, Simonsick EM, Newman AB, Nevitt M, Harris TB. Relationship of interleukin-6 and tumor necrosis factor-alpha with muscle mass and muscle strength in elderly men and women: the Health ABC Study. J Gerontol A Biol Sci Med Sci. 2002 May;57(5):M326-32. doi: 10.1093/gerona/57.5.m326. PMID 11983728
- [Background] Kyle UG, Bosaeus I, De Lorenzo AD, Deurenberg P, Elia M, Gomez JM, Heitmann BL, Kent-Smith L, Melchior JC, Pirlich M, Scharfetter H, Schols AM, Pichard C; Composition of the ESPEN Working Group. Bioelectrical impedance analysis--part I: review of principles and methods. Clin Nutr. 2004 Oct;23(5):1226-43. doi: 10.1016/j.clnu.2004.06.004. PMID 15380917
- [Background] Han CW, Lee EJ, Iwaya T, Kataoka H, Kohzuki M. Development of the Korean version of Short-Form 36-Item Health Survey: health related QOL of healthy elderly people and elderly patients in Korea. Tohoku J Exp Med. 2004 Jul;203(3):189-94. doi: 10.1620/tjem.203.189. PMID 15240928
- [Background] Yun YH, Park YS, Lee ES, Bang SM, Heo DS, Park SY, You CH, West K. Validation of the Korean version of the EORTC QLQ-C30. Qual Life Res. 2004 May;13(4):863-8. doi: 10.1023/B:QURE.0000021692.81214.70. PMID 15129896
- [Background] Lee JH, Lee HJ, Choi YS, Kim TH, Huh YJ, Suh YS, Kong SH, Yang HK. Postoperative Quality of Life after Total Gastrectomy Compared with Partial Gastrectomy: Longitudinal Evaluation by European Organization for Research and Treatment of Cancer-OG25 and STO22. J Gastric Cancer. 2016 Dec;16(4):230-239. doi: 10.5230/jgc.2016.16.4.230. Epub 2016 Dec 20. PMID 28053809
- [Result] Svedlund J, Sullivan M, Liedman B, Lundell L. Long term consequences of gastrectomy for patient's quality of life: the impact of reconstructive techniques. Am J Gastroenterol. 1999 Feb;94(2):438-45. doi: 10.1111/j.1572-0241.1999.874_c.x. PMID 10022643